CLINICAL TRIAL: NCT03561831
Title: Evaluation the Effects of Anaesthetic Agents on Endoplasmic Reticulum Stress During Cancer Surgery
Brief Title: Effect of Anaesthesia on ER Stress in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KUH1160108
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Endoplasmic Reticulum Stress
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): patients who anesthesized by propofol
  Interventions: Drug: Propofol
- sevoflurane group (Active Comparator): patients who anesthesized by sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — propofol based anesthesia
  Arms: propofol group
Drug: Sevoflurane — sevoflurane based anesthesia
  Arms: sevoflurane group

SUMMARY:
Investigate the change in endoplasmic reticulum stress after cancer surgery according to different anaesthetics including propofol and sevoflurane.

DETAILED DESCRIPTION:
We hypothesize propofol and sevoflurane based anesthesia would show different pattern of endoplasmic reticulum stress after cancer surgery in patients with cancer

ELIGIBILITY:
Inclusion Criteria:

- patients with cancer

Exclusion Criteria:

* age under 19 years old
* allergy history to propofol or sevoflurane
* history of previous cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Change in endoplasmic reticulum stress | baseline, postoperative 1 hours and 24 hours
  Change in endoplasmic reticulum stress

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, Professor, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No